CLINICAL TRIAL: NCT03806777
Title: Intra-nasal Dexmedetomidine for Children Undergoing MRI Imaging
Acronym: DexmedMRI
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of British Columbia (Other)
Collaborators: British Columbia Children's Hospital (Other)
Responsible Party: Principal Investigator, Mark Ansermino, Associate Professor, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: H18-02794
Record Dates: First submitted 2019-01-14; First posted 2019-01-16 (Actual); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: MRI Sedation
Keywords: dexmedetomidine
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: Dose finding
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Intra-nasal dexmedetomidine (Experimental): A single dose of dexmedetomidine, determined by a biased coin algorithm (min: 1 mcg/kg; max: 4 mcg/kg or 200mcg), will be delivered intranasally 45min before an MRI scan.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — Highly selective alpha-2 adrenergic agonist with sedative properties.
  Other Names: Precedex

SUMMARY:
This study aims to assess the use of intranasal dexmedetomidine (IN-dex) as a sole agent in aiding the successful completion of a MRI scans in children. Dexmedetomidine, a routinely used anesthetic agent in our institution, has many benefits including sedation with neuro-protective and respiratory sparing features. We will test its effectiveness in completing MRI scans in children that would otherwise be given a full general anesthetic.

DETAILED DESCRIPTION:
Purpose:

To assess the use of IN-dex as a sole agent in aiding the successful completion of a MRI scan in children.

Hypothesis:

We hypothesize that the optimal dose for IN-dex to produce appropriate sedation for MRI will be between 1 and 3 mcg/kg. We also hypothesize that this dose will be lower in the older age group.

Justification:

The dose required for IN-dex to enable safe sedation for MRI scanning as a sole agent is undetermined at present. This study will enable us to find the optimal dose for effective sedation for MRI scanning in a range of age groups. This will avoid the need for propofol and remifentanil general anesthesia (that is the current standard of care) in this group of patients. Our motivation for avoiding general anesthesia is that there is ongoing concern that general anesthesia causes long term neurocognitive effects in children. Finally, identifying a safe yet effective dose of IN-dex, which can be nurse-administered, will also allow us to improve access to MRI scans that are limited by the access to general anesthesia.

Objectives:

1. To determine the dose of IN-dex that, when used as a sole agent, produces minimal to moderate sedation that is adequate for successful completion of MRI in children with >90% effectiveness.
2. To explore the logistics of a nurse-administered sedation protocol to increase access to the MRI.

Research Design:

We propose a dose finding study of IN-dex using the biased coin design (BCD) method in three different age groups (3 to <8 years, 8 to <12 years, 12 to <19 years). The study specific interventions will include identification of children appropriate for the study following detailed assessment using a scoring system developed by our Child Life specialists for use at their MRI preparation session.

Statistical Analysis:

The dose of IN-Dex that produces mild to moderate sedation in 90% of subjects will be calculated using the pooled adjacent violators algorithm (PAVA) and bootstrap methods will be used to calculate the 95% confidence limits.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1 or 2
* Scheduled for elective MRI scan on the general anesthesia list
* Child Life MRI simulation score of 6-10 (Figure 1)
* Age 3 - 18

Exclusion Criteria:

* Taking existing opioid, sedative, or cannabinoid medication
* Severe learning disability defined as the inability to follow simple commands
* Severe Cardiac disease
* Chronic hypertension
* Allergy to dexmedetomidine
* Nasal anatomical abnormality
* Known or anticipated difficult airway

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 180 (Estimated)
Dates: Start 2019-02 (Estimated); Primary Completion 2020-03 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Dose | Immediately after completion of the MRI scan.
  The intranasal dexmedetomidine dose in mcg/kg that produces successful completion of MRI scan with acceptable MRI image quality in 90% of individuals (ED 90).

SECONDARY OUTCOMES:
Uninterrupted scans | Immediately after completion of the MRI scan.
  Total number of scans that were able to be completed without interruptions
Respirator support | During MRI scan
  Total number of occurrences of respiratory support
Adverse events | During MRI scan
  Occurrence of haemodynamic disturbance (bradycardia: absolute heart rate ≤ 40 bpm, hypertension: relative mean arterial pressure ≥ 50% baseline, hypotension: relative mean arterial pressure ≤ 50% baseline)
modified Yale Preoperative Anxiety Scale (mYPAS) | Immediately before administration of intranasal dexmedetomidine
  Pre-procedure mYPAS score. The scale is a total summed score (4-22) of 5 areas; Activity (1-4), Vocalizations (1-6), Emotional expressivity (1-4), state of apparent arousal (1-4), and use of parents (1-4). A lower score represents a lower level of anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Ansermino, FRCA, Principal Investigator — BC Children's Hospital, Department of Anesthesia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Pediatric Anesthesia Research Team website — http://part.bcchr.ca